CLINICAL TRIAL: NCT03569800
Title: Evaluation of the Clinical and Biological Consequences of Levothyrox® Formula Modification
Acronym: FORTHYROX
Status: Terminated | Type: Observational
Why Stopped: investigator's decision : recruitment difficulties and lack of interest in the remote study of the crisis Levothyrox
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18008J; 2018-A00554-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Thyroid Disorder
Keywords: Levothyrox®; thyroid hormones; bioequivalent
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self completed questionnaire — self completed questionnaire

SUMMARY:
The purpose of this study is to determine whether the recent excipient modification of Levothyrox® in France for a bioequivalent formula has clinical and biological consequence for the patients. The investigators also plan to describe the patient journey in terms of levothyroxine based drugs since this formula modification of Levothyrox®.

DETAILED DESCRIPTION:
Levothyrox® is a levothyroxine based drug marketed in France in order to substitute a lack of thyroid hormones. Because of a lack of stability during time and because of wide inter-batch variability in terms of active molecule, the National Agency of Safety of Medicaments (ANSM) ask to the market authorization holder to develop a new formula without lactose. This new formula, which has been proven to be bioequivalent has been marketed since march 2017 in France. Some patients were predicted to have their thyroid function imbalance because of this modification. The purpose of the study is to analyse, on the patients treated by Levothyroxine® in how many patients this modification has clinical and biological consequences.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid disorder treated by Levothyroxine
* Age over 18 year old
* TSH plasma level within the 12 months before formulation modification
* TSH plasma level within the 6 months after formulation modification

Exclusion Criteria:

- Thyroid dysfunction (hypo or hyperthyroidism) despite Levothyroxine treatment, ie TSH plasma level out of normal range within the 6 months before formula modification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population refers to outpatients with a thyroid disorder who consult at the Endocrinology department of Hopitaux Universitaires Paris Centre
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Number of abnormal Thyroid Stimulating Hormone (TSH) level after change of levothyrox formulation | 1 day
  Evaluated with a self completed questionnaire

SECONDARY OUTCOMES:
Number of patients treated with new formulation of levothyrox | 1 day
  Evaluated with a self completed questionnaire
Difference betweenTSH plasma levels before and after formulation change | 1 day
  Evaluated with a self completed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: lionel Groussin, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpitaux Universitaires Paris Centre, Paris, France